CLINICAL TRIAL: NCT03182361
Title: Implant Survival and Peri-abutment Tissue Reactions of Extra-oral Implants: An Interventional Study of 10 Patients
Brief Title: Implant Survival and Peri-abutment Tissue Reactions of Extra-oral Implants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: BioComp Industries bv (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/0282; B670201731744 (Other: Registration of studies Belgium)
Record Dates: First submitted 2017-05-02; First posted 2017-06-09 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Maxillofacial Prosthesis Implantation; Extra-oral Implants; Extra-oral Prosthesis; Prostheses and Implants
Keywords: Auricular, nasal, orbital, extraoral prostheses, extraoral implants, peri-implant reactions, Holgers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Everybody enrolled in the study will receive BioComp Industries cranio-maxillo-facial (CMF) screw implants
  Interventions: Device: Implantation of BioComp Industries cranio-maxillo-facial (CMF) screw implants

INTERVENTIONS:
Device: Implantation of BioComp Industries cranio-maxillo-facial (CMF) screw implants — Placement of BioComp Industries extraoral screw implants with diameters 3.4mm or 4mm and lengths 3.4mm or 4mm in temporal, nasal or orbital bone
  Other Names: EO-1110-34VD04; EO-1110-40VD03; EO-1110-40VD04

SUMMARY:
Patients with craniofacial defects caused by oncologic resection, traumatic events or congenital etiologies suffer from esthetic, functional and psychological problems. Auricular, nasal and orbital defects can be reconstructed with implant retained extra-oral prosthesis. The goal of this study is to evaluate implant survival in temporal, maxillary and orbital bone, and peri-implant tissue reactions using a new implant system developed by BioComp Industries.

DETAILED DESCRIPTION:
Protocol:

1. Planning The ideal size and location of the implants is based on pre-operative CT or CBCT scan followed by analysis using romexis planning software.

   In normal circumstances, without bone limitations, the number and location of the implants will be planned as mentioned below:
   * Left auricular region: 2 implants placed on position 4h and 1h30 in the temporal/mastoid bone. If necessary, 3 implants are placed on positions 1h30, 3h and 4h30. The inter implant distance is 20mm.
   * Right auricular region: 2 implants placed on position 8h and 10h30 in the temporal/mastoid bone. If necessary, 3 implants are placed on positions 10h30, 9h and 7h30. The inter implant distance is 20mm.
   * Nasal region: 2 implants placed in the lateral parts of the piriform aperture of the maxilla, as far away from the spina nasalis anterior as possible. If necessary a third implant will be placed in the glabella.
   * Left orbital region: 2-4 implants are placed in the supra-orbital, lateral and/or infra-orbital rim on positions 1h, 2h, 3h en 5h.
   * Right orbital region: 2-4 implants are placed in the supra-orbital, lateral and/or infra-orbital rim on positions 11h, 10h, 9h en 7h.

   If for some reason there is insufficient bone in the above mentioned areas, the position of the implants will be minimally adjusted in order to secure good osseointegration. Neuronavigation will be used for cases with limited bone volume.
2. Flap design During surgery the first step is the creation of a skin flap or resection of a tumor, exposing the area for implantation.
3. Implantation The implantation protocol as described by BioComp Industries will be used. Each drilling procedure is executed by 1800-2000rpm with water cooling.

   * Defining the implant location with the 2,45mm diameter round bur.
   * Preparation of the implant site with the implant drills, length and diameter of the drill is dependent on the length and diameter of the implant. Drilling protocol will always start with the smallest and shortest drill and gradually expanded, corresponding to the size of the implants.
   * Placement of the implant without water cooling at 15rpm and maximal torque of 52Ncm. If necessary the implant will be inserted manually.

   For auricular, orbital and nasal defects with sufficient bone volume (>=3mm) and good bone quality, a percutaneous healing abutment with torque 20-25 ncm will be placed immediately after insertion of the implant (=one-stage protocol). Soft tissues in an area of 15-20mm surrounding the implant will be reduced to 1mm thickness.

   In all other circumstances, the implant will be protected by means of a cover screw and reburied under the skin for a 3 month osseointegration period (=two-stage protocol). After 3 months the implants are exposed, percutaneous healing abutments placed and the surrounding soft tissues reduced to 1mm thickness.

   In the case of large resections where no viable skin is left, a split thickness skin graft from the upper thigh will be used.

   Finally, a healing cap surrounding the healing abutments is placed to ensure strong bone-skin contact around the implant. This healing cap will be fixated by a fixation screw, torqued at 15 Ncm.
4. Clinical measurements:

   The stability of the implants will be measured at the time of abutment placement, 1 or 2 weeks, 1 month, 3 months, 6 months and yearly until the end of the study by resonance frequency analysis (RFA), using the Osstell idx system.

   At the same time periods the peri-abutment tissue will be evaluated according to the Holgers criteria.

   Once all implants have reached a stability measurement of 50 ISQ, the patient will be sent to the anaplastologist for prosthesis treatment.

   In case one or more of the implants fail during the study period, the implant will be removed and replaced by a new implant. The protocol will restart for the newly placed implant.
5. Radiological measurements:

The bone level around the implants will be measured at 1 or 2 weeks after implant placement and 1 year after implant placement. Radiological imaging will be performed using a cone beam computed tomography device (planmeca promax 3d max) or CT scan, dependent on primary imaging in order to allow comparison between both images.

ELIGIBILITY:
Inclusion Criteria:

* All patients with auricular, nasal, orbital defects caused by congenital, traumatic, oncologic or infectious etiologies
* Adults (>18yr)

Exclusion Criteria:

* Children
* Implant placement for bone anchored hearing aid (BAHA)
* Implant placement for oral rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Implant survival | 1 year
  Implant stability measurement with Osstell IDX system
Peri-implant tissue reaction | 1 year
  Measurement of peri-implant pockets and soft tissue according to Holgers criteria

SECONDARY OUTCOMES:
Bone level | 1-2 weeks post-operative, 1 year
  Bone level measurement using CBCT or CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Vermeersch, MD, PhD, Principal Investigator — Em. Professor
Locations (1):
- University Hospital, Ghent, Oost-Vlaanderen, Belgium